CLINICAL TRIAL: NCT04992598
Title: Hypnosis to Reduce Pain and Drugs for Shoulder Dislocation Management in the Emergency Department
Brief Title: Hypnosis to Reduce Pain and Drugs for Shoulder Dislocation Management
Acronym: HYPSEM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of the study coordinating investigator
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-02-CHRMT
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Dislocation
Keywords: Hypnosis
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis group (Experimental)
  Interventions: Other: Hypnosis session; Procedure: Reduction
- Control group (Placebo Comparator)
  Interventions: Procedure: Reduction

INTERVENTIONS:
Other: Hypnosis session — Hypnosis session will precede therapeutic strategies and reduction
  Arms: Hypnosis group
Procedure: Reduction — All dislocation would be reduced Under adequate analgesia and sufficient sedation. All methods for reduction can be used.

SUMMARY:
The effectiveness of hypnosis for reducing pain was evaluated in various medical specialities. However, only few studies have demonstrated the efficacy of hypnosis for the management of pain in the emergency medicine.

Anteromedial dislocation is a very common Reason for admission in emergency department. Many methods for reduction have been described but there is no consensus on the optimum technique or sedation procedures.

Some pain medication and tranquilizers used during a shoulder dislocation management include hemodynamic, respiratory and behavioral adverse effects with the requirement of strengthened surveillance.

Hypnosis could provide to reduce sedative and analgesic use during the reduction of anteromedial dislocation.

The main objective of this study is to evaluate the efficacy of a hypnosis session for reducing the consumption of analgesic in patient throughout a reduction of shoulder dislocation.

The investigators also examine the effect of hypnosis on hemodynamic parameters, patient's pain, patient and practitioner satisfaction, sedative consumption, number of attempts for reduction and length of stay in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over,
* Checked into ED for an anterior shoulder dislocation suspected by clinical examination and confirmed by radiography,
* Had given oral consent to participate in the study
* Are affiliated or be a recipient of a social security plan.
* A staff member (nurse, nurse's aide, or physician) trained in hypnosis is available at the patient admission time.

Exclusion Criteria:

* Patient showing up with a shoulder fracture on x-ray.
* Patient presenting a shoulder prosthesis.
* Patient with recurrent dislocations.
* Patient who does not speak or understand French language.
* Patient with cognitive dysfunction.
* Patient with a psychiatric history of psychosis.
* Patient who is deaf or hard of hearing.
* Patient under legal protection (guardianship, curatorship).
* Pregnant women
* Patient who already benefited of a pre-hospital reduction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | Day 1
  Calculated as the equal dose of morphine

SECONDARY OUTCOMES:
Dose of sedative drug | Day 1
  Dose of sedative drug
Patients'satisfaction | Day 1
  Patients'satisfaction was assessed with a Likert scale after reduction. The satisfaction was scored on 5-point Likert scale, ranging from 1 to 5 (with 1=excellent and 5=catastrophic).
Practitioners'satisfaction | Day 1
  Practitioners'satisfaction was assessed with a Likert scale after reduction. The satisfaction was scored on 5-point Likert scale, ranging from 1 to 5 ( with 1=excellent and 5=catastrophic).
Number of attempts for reduction | Day 1
  Number of attempts for reduction
Length of stay | Day 1
  Length of stay in the emergency department
Method use for reduction | Day 1
  Method use for reduction
Adverse events | Day 1
  number of adverse events

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHR Fleyriat- Hôpital de Bourg en Bresse, Bourg-en-Bresse, Ain
  - Centre Hospitalier Lucien Hussel, Vienne, Isère
  - CHR Metz Thionville, Metz, Moselle
  - Hôpital Robert Pax, Sarreguemines, Moselle
  - Centre Hospitalier Saint Luc Saint Joseph, Lyon, Rhône
  - Groupement hospitalier Sud-Hôpital Lyon Sud, Lyon, Rhône
  - Hôpital Nord-Ouest Villefranche sur Saône, Villefranche-sur-Saône, Rhône

REFERENCES:
- [Derived] Tinelli M, Guler N, Goetz C, Aim P, Marchionni S, Ouamara N, Cipolat L, Demarquet M, Seris E, Moreau A, Durand G, Douplat M, Lavignon JP, Hingray C, Abensur Vuillaume L. Study protocol: hypnosis versus standard care for shoulder dislocation reduction in the emergency department - a multicentre, randomised, controlled study protocol. BMJ Open. 2022 Dec 7;12(12):e062278. doi: 10.1136/bmjopen-2022-062278. PMID 36600368